CLINICAL TRIAL: NCT05822310
Title: Comparison of Femoral and Obturatory Nerve Joint Branches Conventional Radiofrequency Thermocoagulation ,Intraarticular Steroid Injection and Pericapsular Nerve Group (PENG) Block in Chronic Hip Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, SINEM SARI, Associate professor, Aydin Adnan Menderes University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2022/07
Record Dates: First submitted 2023-01-19; First posted 2023-04-20 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Chronic Hip Pain
Keywords: femoral and obturatuar nerve; chronic hip pain; Radiofrequency thermocoagulation; intraartıcular steroid injection; pericapsular nerve group (PENG) block
MeSH Terms: conditions — Bites and Stings | interventions — Dental Occlusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- radiofrequency thermocoagulation to the articular branches of the femoral and obturatory nerves (Experimental): radiofrequency thermocoagulation to the articular branches of the femoral and obturatory nerves applied
  Interventions: Procedure: radiofrequency thermocoagulation to the articular branches of the femoral and obturatory nerves
- intraairticular steroid injection (Active Comparator): intraairticular steroid injection applied
  Interventions: Procedure: intraairticular steroid injection
- pericapsular nerve group (PENG) block (Active Comparator): pericapsular nerve group (PENG) block applied
  Interventions: Procedure: pericapsular nerve group (PENG) block

INTERVENTIONS:
Procedure: radiofrequency thermocoagulation to the articular branches of the femoral and obturatory nerves — Patients are operated under sedation in the operating room. C-arm fluoroscopy device is used for imaging purposes for radiofrequency thermocoagulation process. In order to prevent vascular injury, the needle is advanced under the guidance of ultrasonography. There are target points determined in fluoroscopy for the femoral nerve and the obturatory nerve. Before the thermocoagulation procedure, local anesthetic and steroid are injected into each of the target points.
  Arms: radiofrequency thermocoagulation to the articular branches of the femoral and obturatory nerves
Procedure: intraairticular steroid injection — The patients were placed in the supine position in the operating room. The patient was stained sterile with povidone iodide. The femoral neck was detected under ultrasonography and the joint capsule was entered with a 22G 9 cm spinal needle. Then, 5 cc bupivacaine and 5 mg betamethasone were given and the procedure was terminated.
  Arms: intraairticular steroid injection
Procedure: pericapsular nerve group (PENG) block — The patients were placed in the supine position in the operating room. The patient was stained sterile with povidone iodide. The high-frequency linear ultrasonography probe was placed on the anterior superior iliacspina (ASIS). Later, the anterior inferior iliac spine (AIIS) was detected by descending caudally. Afterwards, the probe was brought to the oblique position and AIIS, iliopubikeminence, psoas muscle and tendon were seen. Using a 22G 90-mm Quinckespinal needle, the tendon of the iliopsoas muscle was entered in the lateral-medial direction in the in-plane plane and bone contact was achieved. After negative aspiration, 15 ml of 0.5% bupivacaine were administered by seeing the appropriate drug distribution.
  Arms: pericapsular nerve group (PENG) block

SUMMARY:
In this study ,the investigators aimed to show the decrease in pain levels and the effect on quality of life of patients who underwent chronic hip painRFT , intraartıcular steroid injection and Peng block.

DETAILED DESCRIPTION:
Hip pain is a common medical condition with increasing age.The effectiveness of conservative methods used in hip pain is limited.Since the lifespan of prostheses used in hip surgery is limited, new methods are needed in the treatment of pain.The anterior sensory innervation of the hip joint is provided by the articular branches of the femoral and obturatory nerve. Today, the most commonly used techniques for hip pain are corticosteroid administration into the hip joint, pericapsular nerve group (PENG) block application, and radiofrequency thermocoagulation to the articular branches of the femoral and obturatory nerves. The aim of this study is to compare the effects of these three procedures in hip pain.

ELIGIBILITY:
Inclusion Criteria:

1. be over 18 years old
2. Written consent has been obtained
3. Those with chronic hip pain for more than 3 weeks

Exclusion Criteria:

1. Major psychiatric illness
2. The patient has lumbar compression pain or referred pain
3. Patients using anticoagulant agents
4. Patients with infection in the area to be treated
5. Those who are allergic to local anesthetics
6. Those who are allergic to betamethasone
7. Pregnancy
8. Patients who underwent hip surgery during the 3-month follow-up period during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-04-15 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
NRS(Numerating Rating Scale) for chronic pain | preoperative
  İt is a pain intensity determination system based on the system where there person tells a point between 0=(no pain) 10=( unbearable pain) and to describe their pain
NRS(Numerating Rating Scale) for chronic pain | Postoperative first month
  İt is a pain intensity determination system based on the system where there person tells a point between 0=(no pain) 10=( unbearable pain) and to describe their pain
NRS(Numerating Rating Scale) for chronic pain | Postoperative third month
  İt is a pain intensity determination system based on the system where there person tells a point between 0=(no pain) 10=( unbearable pain) and to describe their pain

SECONDARY OUTCOMES:
WOMAC (Western OntarioandMcMasterUniversitiesArthritisIndex ) | Preoperative
  It includes 24 questions under three sub-headings as pain, stiffness and physical function. Each question was scored according to the Likert scale as 0=absent, 1=mild, 2=moderate, 3=severe, 4=very severe.minimum score is 0=good maximum score is 96 = bad functional capacity
WOMAC (Western OntarioandMcMasterUniversitiesArthritisIndex ) | Postoperative first month
  It includes 24 questions under three sub-headings as pain, stiffness and physical function. Each question was scored according to the Likert scale as 0=absent, 1=mild, 2=moderate, 3=severe, 4=very severe.minimum score is 0=good maximum score is 96 = bad functional capacity
WOMAC (Western OntarioandMcMasterUniversitiesArthritisIndex ) | Postoperative third month
  It includes 24 questions under three sub-headings as pain, stiffness and physical function. Each question was scored according to the Likert scale as 0=absent, 1=mild, 2=moderate, 3=severe, 4=very severe.minimum score is 0=good maximum score is 96 = bad functional capacity

OTHER OUTCOMES:
NRS(Numerating Rating Scale) for acute pain | postoperative second hour
  İt is a pain intensity determination system based on the system where there person tells a point between 0=(no pain) 10=( unbearable pain) and to describe their pain

CONTACTS AND LOCATIONS:
Locations (1):
- Adnan Menderes University Faculty of Medicine, Aydin, Turkey (Türkiye)